CLINICAL TRIAL: NCT06527495
Title: Clinical Pharmacogenetic Study of the Efficacy and Safety of Sorafenib in Egyptian Patients With Hepatocellular Carcinoma
Brief Title: Clinical Pharmacogenetic Study of Sorafenib in Egyptian Patients With Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Nazih, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00470/2023
Record Dates: First submitted 2024-07-13; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: HCC; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sorafenib (Experimental): Sorafenib 200 - 400 mg twice daily
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Sorafenib Tablets (200 -400 mg) twice daily

SUMMARY:
The current study will aim to maximize the therapeutic effect and to minimize the adverse effects of sorafenib in HCC through pharmacogenomic analysis of VEGFA and KDR genetic polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* Age of all studied subjects ≥ 18 years old
* All patients with hepatocellular carcinoma will be included in group I.
* Patients not treated with systemic TKIs

Exclusion Criteria:

* Patients presented with liver tumors other than HCC.
* Patients with Child-Pugh grade C for liver function.
* Patients with other malignancies.
* Patients with chronic inflammatory disorders.
* Patients with severe organ dysfunction such as heart, lung, and kidney.
* Patients who cannot tolerate or are allergic to sorafenib.
* Patients with severe coagulation dysfunction were uncorrectable.
* Age less than 18 years old.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Vascular Endothelial Growth Factor A (VEGFA) genotyping | At Baseline, 3 month, and 6 month after treatment.
  Genetic polymorphism of VEGFA
Kinase insert domain receptor (KDR) genotyping | At Baseline, 3 month, and 6 months after treatment.
  Genetic polymorphism of KDR

SECONDARY OUTCOMES:
Tumor markers | At Baseline, 3 month, and 6 month after treatment.
  Determination of serum Alpha-Fetoprotein, AFP-L3
Complete blood culture | At Baseline 3 month, and 6 months after treatment.
  Determination of hemoglobin concentration
Kidney function tests | At Baseline 3 month, and 6 months after treatment.
  Determination of Serum creatinine concentration
Liver function tests. | At Baseline 3 month, and 6 months after treatment.
  Determine serum level of ALT and AST
Safety outcome | At Baseline, 3 month, and 6 months after treatment.
  Incidence of side effects such as (diarrhea, anorexia, nausea, vomiting, hand and foot syndrome)

CONTACTS AND LOCATIONS:
Locations (1):
- NLI, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No